## Johnson & Johnson Vision

## STATISTICAL ANALYSIS PLAN

#### **Protocol** CR-6400

Clinical Evaluation of a Daily Wear Reusable Multifocal Optical Design in a Presbyopic Population

## JJV Investigational senofilcon A Multifocal Contact Lens

Version: 1.0

Date: 3 November 2020

**Compliance:** The study described in this document was performed according to the principles of Good Clinical Practice (GCP).

## **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this document and the attachments.

| Author | | |
|----------|-----------------------------------------|------------------|
| | | DATE:03 NOV 2020 |
| Reviewer | | |
| | | DATE:03 NOV 2020 |
| Approver | | |
| | Name: Thomas R Karkkainen, OD, MS, FAAO | DATE:03 NOV 2020 |

# **TABLE OF CONTENTS**

| AU1 | THORIZED SIGNATURES | 2 |
|---|---|---|
| TAE | BLE OF CONTENTS | 3 |
| AMI | ENDMENT HISTORY | 5 |
| ABE | BREVIATIONS | 5 |
| 1. | INTRODUCTION | |
| 2. | STUDY OBJECTIVES | |
| 3. | STUDY DESIGN | |
| 3.1. | Overview | |
| 3.2.<br>3.3. | Test Articles Targeted Study Population and Sample Size | |
| 3.4. | Test Article Allocation and Masking | |
| 3.5. | Time and Event Schedule | |
| <b>4.</b><br>4.1. | STUDY ENDPOINTSSecondary Endpoints | |
| 4. 1.<br>4.2. | Other Endpoints | |
| | ' | |
| 5. | STATISTICAL HYPOTHESES FOR STUDY OBJECTIVES | |
| 5.1. | Primary Hypotheses | |
| 5.2.<br>5.3. | Secondary Hypotheses Other Hypotheses | |
| J.J. | | |
| 6. | ANALYSIS SETS | |
| 6.1. | All Enrolled | |
| 6.2.<br>6.3. | Intent-to-Treat (ITT) | |
| 6.4. | Safety Population<br>Per-Protocol (PP) | |
| 7. | DEFINITIONS AND DERIVED VARIABLES | |
| 7.1. | Age | |
| 7.2.<br>7.3. | Visit Windows | |
| 7.3.<br>7.4. | Average daily wear time (in Hours) | |
| 8. | GENERAL STATISTICAL CONSIDERATIONS | |
| 8.1.<br>8.2. | Statistical Software | |
| 8.2.<br>8.3. | Summary StatisticsReporting Numerical Values | |
| 6.3.<br>8.4. | Sample Size Justification | |
| 8.5 | Statistical Significance Level | 15 |

| 8.6. | Handling of Missing Data and Drop-outs | . 15 |
|---|---|---|
| 9. II | NTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | . 15 |
| 10. \$ 10.1. 10.2. 10.3. 10.4. 10.5. 10.6. | Treatment Compliance and Extent of Exposure Prior and Concomitant Medications | . 15<br>. 16<br>. 16<br>. 16<br>. 16 |
| 11.1.<br>11.2. | Primary AnalysisSecondary Analysis | . 17<br>. 22 |
| | Contact lens Corrected Visual Acuity Reasons for Discontinuation Unscheduled Lens Replacement Physical Examination Findings Clinical Laboratory Tests | . 23<br>. 23<br>. 23<br>. 23<br>. 24<br>. 24 |
| | REFERENCES | |
| 14.1.<br>14.2. | APPENDICES Time and Event Schedule Statistical Analysis Code | . 27<br>. 30 |

# AMENDMENT HISTORY

| Version Number | Revision Date<br>(DD/MM/YYYY) | Reasons for Revision |
|----------------|-------------------------------|----------------------|
| 1.0 | 03 November 2020 | Original |

## **ABBREVIATIONS**

| | TANK THE REPORT OF THE PERSON |
|---|---|
| AE | adverse event |
| CLVA | Contact Lens Visual Acuity |
| CrI | Credible interval |
| CRF | case report form |
| CSR | Clinical Study Report |
| DMC | Data Monitoring Committee |
| eCRF | electronic case report form |
| FDA | Food and Drug Administration |
| HLHC | High Luminance High Contrast |
| ICH | International Conference on Harmonization |
| ITT | Intent-to-Treat |
| IVRS | interactive voice response system |
| LOCF | last observation carried forward |
| PI | principal investigator |
| SAE | serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | standard deviation |
| VP | Visual Performance |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the analyses and data presentations for protocol CR-6400 Version 4.0.

This document will serve as the final guidance for all the statistical analysis for this study and will supersede the Statistical Method section in the protocol if there are any discrepancies. Any deviation from the analysis plan will be documented as such in the clinical study report.

#### 2. STUDY OBJECTIVES

## Primary Objective:

The primary purpose of this study is to demonstrate that the Multifocal Test lens made with senofilcon A material made from the Flexible Manufacturing Platform (FMP), in its final lens design FAL100, FAL101 and FAL102 (low, mid and high ADD respectively) meets the design validation requirements for CLUE overall quality of vision scores, logMAR visual acuity, ocular physiology and lens fit acceptance.

## Secondary Objective:

The secondary objective is to evaluate the number of lenses needed to optimize the subject's vision.

#### 3. STUDY DESIGN

#### 3.1. Overview

The clinical study is a bilateral, single-masked (partial), single-arm, clinical trial. A total of approximately 60 eligible subjects (30 myopes and 30 Hyperopes) will be targeted to complete the study.

The study begins with an initial visit, Visit 1 (Day 0), if a subject is found to meet all eligibility criteria, they will be fit with the study lens, in both eyes; otherwise the subject will be deemed ineligible and classified as a screen failure.

If a subject is dispensed lenses at the initial visit, then two additional visits will be conducted. Visit 2 will occur  $3 \pm 1$  days after Visit 1. At Visit 2 subjects will undergo lens optimization if the subject reports unsatisfactory vision or is unable to obtain 20/30 binocular distance visual acuity with the study lenses. Subjects will return for Visit 3 (Final Evaluation) after  $12\pm 2$  days. At the final visit, subjects will undergo subjective and objective assessments of vision.

Subjects will be advised to wear the study lenses every day while they are in the study for a minimum of 6 hours per day. The study lens will be replaced at the optimization visit. However, lost or damaged lenses maybe replaced when necessary. Unscheduled visit may be conducted.

#### 3.2. Test Articles

Table 1: Test article labels

| Test Article | Label |
|---------------------------------------------|-------|
| JJV Investigational Multifocal Contact Lens | Test |
| ACUVUE OASYS® with HYDRACLEAR® PLUS Sphere* | Test |
| All Test Articles | Total |

<sup>\*</sup>Note: The spherical test lens (JJV Investigational Multifocal Contact Lens) is used in the troubleshooting steps only for low ADD subjects who have reported a distance vision complaint.

# 3.3. Targeted Study Population and Sample Size

Approximately 80 subjects will be enrolled to ensure that 60 subjects will complete the study (30 myopes and 30 hyperopes). Enrolled subjects will be habitual wearers of soft contact lenses. All subjects will be at least 40 years of age and not older than 70 years of age at the time of enrolment. Eligible presbyopes will be those that wear an a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (CR-6400 Protocol Version 4.0, Appendix E).

Table 2: Planned Enrollment Strategy by Strata and Site

| | Myopes | Hyperopes | Total |
|----------------------------------------------|--------|-----------|-------|
| Enrolled | 40 | 40 | 80 |
| Randomized | 30 | 30 | 60 |
| Number of enrolled per site (min-max) Target | 2-6 | 2-6 | |

## 3.4. Test Article Allocation and Masking

The study lenses will be worn in a bilateral fashion using a single-arm design. Due to the nature of the design no randomization is required.

This is a single arm study and all subjects will be assigned to the same study lens. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

## 3.5. Time and Event Schedule

See Appendix 14.1 for details regarding the Time and Events Schedule.

# 4. STUDY ENDPOINTS

Primary Efficacy Endpoints:

### **CLUE Overall Quality of Vision**

Overall comfort scores will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>)<sup>1</sup> questionnaire after approximately 2 weeks of lens wear. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.

## Visual Acuity (logMAR)

Multiple assessments of binocular and monocular visual acuity will be made during the study, but the binocular measurements made after approximately 2 weeks of lens wear using high contrast letters in bright illuminance conditions will be the primary endpoint. At distance (4 meters), VA is assessed using ETDRS charts; while near (40 cm) and intermediate (64 cm) assessments will be made using reduced Guillon-Poling charts. Visual acuity will be measured using high and low contrast charts in bright illuminance conditions.

Primary Safety Endpoints:

#### Slit Lamp Findings (SLF)

Slit Lamp Findings (Grade 3 or higher) will be assessed for each subject eye at all study visits (schedule and unscheduled). SLFs will be evaluated and classified using the FDA Grading scale rating from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1=trace, Grade 2= mile, Grade 3=moderate and Grade 4= severe). The percentage of eyes with Grade 3 or higher slit lamp findings will be analyzed and will include corneal infiltrates.

### Unacceptable Lens Fit

Unacceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each subject eye. Unacceptable fit is a binary response where Y=1 if lens fit is unacceptable and

Y=0 otherwise. Unacceptable fit was defined as unacceptable if any one of the following criteria:

- limbal exposure at primary gaze or with extreme eye movement;
- edge lift;
- excessive movement in primary up gaze;
- insufficient movement in all three of the following conditions: primary gaze, up gaze, and push up test.

Eyes with multiple unacceptable fitting events was counted only once. See CTP-2008 in Appendix H for additional details regarding lens fit assessments.

# 4.1. Secondary Endpoints

Summary of lenses needed to fit (optimize) the subject's vision

# 4.2. Other Endpoints

- Lens Deposits
- CLUE comfort/handling scores
- GSI Product Performance ratings

### 5. STATISTICAL HYPOTHESES FOR STUDY OBJECTIVES

# 5.1. Primary Hypotheses

All the following co-primary hypotheses must be satisfied in order to meet the study objectives.

#### Primary Hypotheses:

- 1. After approximately 2-weeks of wear, the mean overall quality of vision score of the Test lenses will be statistically better than 40 points for the myope population. This will be recorded by the subject using the CLUE Follow-up Questionnaire.
- 2. After approximately 2-weeks of wear, the mean overall quality of vision score for the Test lenses will be statistically better than 32 points for the hyperope population. This will be recorded by the subject using the CLUE Follow-up Questionnaire.
- 3. After approximately 2-weeks of wear, the mean distance, binocular, high luminance, high contrast logMAR visual acuity score of the Test lens will be statistically lower than 0.10 logMAR.
- 4. After approximately 2-weeks of wear, the mean intermediate, binocular, high luminance, high contrast logMAR visual acuity score of the Test lens will be statistically lower than 0.17 logMAR.
- 5. After approximately 2-weeks of wear the mean near, binocular, high luminance, high contrast logMAR visual acuity score of the Test lens will be statistically lower than 0.17 logMAR.

- 6. When wearing the Test lenses, the proportion (%) of eyes with at least one reported clinically significant slit-lamp finding (Grade 3 or 4) during the post-fit period will be significantly lower than 5%.
- 7. When wearing the Test lenses, the proportion (%) of eyes with an unacceptable fit during the study will be statistically less than 5%.

If all the primary hypotheses are met, the following secondary hypothesis will be tested.

## 5.2. Secondary Hypotheses

1. The proportion of subjects who obtain the optimum lens pair in 4 lenses or less will be at least 90% using a 95% level of confidence.

# 5.3. Other Hypotheses

Not applicable.

#### 6. ANALYSIS SETS

#### 6.1. All Enrolled

The All Enrolled population will include all participants who sign an informed consent.

## 6.2. Intent-to-Treat (ITT)

Intent-to-treat will include all enrolled subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 6.3. Safety Population

All subjects who were administered any test article with at least one observation recorded excluding subjects who dropped out prior administering any test article. Safety analyses will be based on the safety population.

#### 6.4. Per-Protocol (PP)

Per Protocol Analysis set will be the primary analysis population. It will include all subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

The following is a preliminary list of criteria that may disqualify a subject from the Per-Protocol analysis. This list is simply suggestive and is subject to change at the pre-lock review:

#### 7. DEFINITIONS AND DERIVED VARIABLES

## 7.1. Age

Age will be calculated using the Date of Birth (DOB) and the date of the consenting the subject and presented as age at last birthday as an integer.

Age = Integer part of [(Date of Baseline visit – Date of Birth) / 365.25]

#### 7.2. Visit Windows

Table 3: Visit window information

| Scheduled Visit | Time Interval | Time Interval | Target Time |
|-----------------|-------------------|--------------------|-------------|
| Number | (label on output) | (Day) <sup>a</sup> | Point |
| 1 | Screening | 0 | 1 |
| 1 | Baseline | 0 | 1 |
| 2 | 3-Day Follow-up | 2 to 4 | 3 |
| 3 | 2-Week Follow-up | 10 to 14 | 14 |

<sup>&</sup>lt;sup>a</sup> The first treatment day is Day 0.

# 7.3. Average daily wear time (in Hours)

Average daily wear time will be calculated as the number of hours between subjects reported time of insertion and time of removal of the study lenses at screening 3-Day Follow-up and 2-Week Follow-up evaluation.

# 7.4. Definition of Subgroups

Subject will be categorized into either the Hyperope or the Myope group based on the subjects' distance spherical refraction. Subjects who have a negative distance spherical refraction will be categorized as a Myope while subjects who have a positive distance spherical refraction will be categorized as a Hyperope. However, if a subject has positive distance spherical refraction in one eye and plano refraction in the opposite eye then the subject will be categorized as a Hyperope. If the subject has negative distance spherical refraction in one eye and plano refraction in the opposite eye, then the subject will be categorized as a Myope. If the subject has positive distance spherical refraction in one eye and negative distance spherical refraction in the other eye, the eye with the highest absolute power (D) will be used to categorize the subject (i.e. if a subject spherical distance refraction is OD: +0.75, OS: -1.25; then they will be categorized as a Myope. If the subject has equal magnitude of spherical refraction but opposite sign between eyes, the subject will be categorized as a Myope.

#### 8. GENERAL STATISTICAL CONSIDERATIONS

## 8.1. Statistical Software

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC)<sup>2</sup>.

# 8.2. Summary Statistics

Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the efficacy statistical analysis but will be included in the analysis of safety endpoints (slit lamp findings and lens fitting).

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum, and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Safety and efficacy variables will be summarized on both safety and PP populations.

## 8.3. Reporting Numerical Values

Means, medians and confidence/credible intervals will be reported to one decimal place greater than the original data. The standard deviation will be reported to two decimal places greater than the original data. Minimum and maximum will use the same number of decimal places as the original data. P-values greater or equal than 0.0001 will be reported to 4 decimal places; p-values less than 0.0001 will be reported as "<0.0001". All percentages will be reported to one decimal place.

## 8.4. Sample Size Justification

This study was designed and powered to demonstrate that the Multifocal Test lens made with senofilcon A material made from the Flexible Manufacturing Platform (FMP), in its final lens design FAL100, FAL101 and FAL102 (low, mid and high ADD respectively) meets the design validation requirements for the following efficacy and safety endpoints:

- CLUE vision score at 2-week follow-up
- Binocular visual acuity (Distance, Intermediate and Near) at 2-week follow-up
- Proportion of eyes with a significant slit lamp finding (Grade 3 or higher)
- Proportion of eyes with unacceptable lens fitting

The historical data used for the sample size calculation were from 6 JJVC sponsored studies. Table 4 displays the studies, their corresponding study design and the number of subjects enrolled and

completed. The investigational product in all these studies was the multifocal Test lens in its' final design (FAL100, FAL101 and FAL102) made from different manufacturing platforms.

Table 4: Historical Studies Utilized for Sample Size Calculation

| Study | Study Design | Manufacturi<br>ng Platform | #Enrolled | #Completed | Population | SKU |
|---|---|---|---|---|---|---|
| | Crossover | FMP <sup>1</sup> | 46 | 43 | Hyperopes | +1.00 to +4.00 |
| | Crossover | TAM21 <sup>2</sup> | 71 | 61 | Hyperopes | +1.00 to +4.00 |
| | Crossover | TAM21 | 63 | 60 | Myopes | -1.00 to-4.00 |
| | Crossover | SCLM <sup>3</sup> | 45 | 45 | Hyperopes | +1.00 to +4.00 |
| | Parallel | MCLM <sup>4</sup> | 189 | 168 | Myopes | -1.00 to-4.00 |
| | Crossover | SCLM | 40 | 34 | Hyperopes | +1.00 to +4.00 |
| Total | | | 454 | 411 | | |

<sup>&</sup>lt;sup>1</sup>FMP: Flexible Manufacturing Platform

Summaries of efficacy data pooled across all the 6 studies are presented in Table 5. Results showed that near, intermediate and distance VA have similar variation across studies, therefore a 0.11 was utilized for the variation in the power calculation for all positions. Historical data have shown that the average CLUE vision score of hyperopes is lower that of myopes.

Table 5: Descriptive summary of Efficacy Endpoints Period 1 Only - 2-Week Follow-up

| | | | Standard | | |
|---|---|---|---|---|---|
| Endpoint | Mean | Median | Deviation | Minimum | Maximum |
| Distance VA (3m) | -0.077 | -0.100 | 0.1026 | -0.320 | 0.560 |
| Intermediate VA (64cm) | -0.054 | -0.060 | 0.1014 | -0.300 | 0.360 |
| Near VAR (40cm) | 0.077 | 0.060 | 0.1100 | -0.260 | 0.460 |
| Hyperopes' CLUE Vision score | 47.71 | 48.07 | 17.514 | 10.22 | 93.50 |
| Myopes' CLUE Vision score | 56.46 | 53.37 | 19.227 | 21.51 | 108.04 |

The proportion of eyes with Grade 3 or higher SLFs and the proportion of eyes with unacceptable lens fittings pooled across all historical studies is presented in the table below. As shown, there was only 1 unacceptable lens fitting in any of the 6 historical study while there have been 5 eyes with reported Grade 3 or higher SLFs.

Table 6: Descriptive Summary of Safety Endpoints all available Data

| Endpoint | Test |
|---------------------------|---------|
| | n(%) |
| Unacceptable lens fitting | 1 (0.2) |
| SLF Grade 3+ | 5 (1.4) |
| Total Eyes (N) | 350 |
| Total Subjects | 175 |

<sup>%=</sup> nx100/N

<sup>&</sup>lt;sup>2</sup>TAM21: Tokyo Automatic Machinery -3GT (3<sup>rd</sup> Generation Technology) manufacturing line

<sup>&</sup>lt;sup>3</sup>SCLM: Single Cavity Lens Machine <sup>4</sup>MCLM: Multi Cavity Lens Machine

#### Safety Analysis

Our plan for safety analysis is to incorporate historical individual subject data from the 6 studies using power prior distributions in a Bayesian framework (see section 14.5). The level of influence of historical data on current is determined by a discounting factor a constrained between 0 and 1  $(0 \le a_0 \le 1)$ .  $a_0 = 0$  corresponds to no borrowing of the historical data; while  $a_0 = 1$  corresponds to full borrowing (See section 14.5 for more details). For this study we considered a low level of borrowing ranging by 0.1 and 0.30 based on the manufacturing platform where the historical study lens was made from. Table 7 displays the number of subjects and the degrees of borrowing that will be used in the safety analysis. The approved investigational product will be manufactured from the FMP platform; therefore, the borrowing strength is larger to lenses from the FMP platform. Furthermore, the TAM21 platform is considered equivalent with respect to lens performance and lenses from these platforms are given the same borrowing strength as those from the FMP platform. While all historical studies used the lens in its final design, lenses made from the pilot line are only given a borrowing strength of 10%.

Table 7: Degrees of Borrowing Historical Data by Manufacturing Platform

| Manufacturing Platform | Number of Subjects | Level of borrowing $(a_0)$ |
|-------------------------|--------------------|----------------------------|
| FMP | 23 | 0.3 |
| TAM21 | 66 | 0.3 |
| Pilot Line (SCLM, MCLM) | 86 | 0.1 |

We calculated the required sample size with and without borrowing historical data. To achieve a minimum of 80% power with a 2-sided type I error rate of 5%, the required sample size with no borrowing ( $a_0 = 0$ ) was 120 subjects (240 eyes); while the sample size with borrowing was 60 subjects (120 eyes). The sample calculation in each scenario of borrowing was conducted using a Monte Carlo simulation of 1000 trials of samples of size 120 subjects (240 eyes) were drawn from a multivariate binary distribution assuming a compound symmetric (CS) covariance structure between left and right eye from the same subject. Assuming a true proportion of eyes with grade 3 or higher SLFs of p=0.014 and a correlation of  $\rho$ =0.70 between left and right eyes. The same approach was considered for the proportion of eyes with unacceptable fitting assuming a true proportion of eyes with unacceptable fit of p=0.01 and a correlation of  $\rho$ =0.80 between left and right eyes.

The sample size was mainly driven by safety analysis, the power calculation of the efficacy analysis showed that a sample size of 60 subjects is sufficiently large to test the efficacy hypotheses. No borrowing was considered for the primary efficacy analysis. Table 8 summarize the statistical power of a sample size of 60 subjects (120 eyes) for all endpoints.

| | 1 21 | | J |
|---|---|---|---|
| Endpoint | Borrowing | Hypothesis (H <sub>A</sub> ) | Power (%) |
| Grade 3 or Higher SLFs | Yes | $p_t < 0.05$ | 80 |
| Unacceptable lens tit | Yes | $p_t < 0.05$ | 90 |
| VA Distance | No | $\mu_{\rm t}$ < +0.10 | > 99 |
| VA Intermediate | No | $\mu_{\rm t} < +0.17$ | > 99 |
| VA Near | No | $\mu_{\rm t}$ < +0.17 | > 99 |
| CLUE Vision (Hyperopes) | No | $\mu_t \ge 32$ | 99 |
| CLUE Vision (Myopes) | No | $\mu_t \ge 40$ | 99 |

Table 8: Power calculation by endpoint/hypothesis assuming a sample size of 60 subjects

The power calculation of the efficacy analyses (CLUE and VA) was conducted using historical data presented in Table 5 above using PROC POWER for one sample means test for equivalence to test each hypothesis.

The plan is to enroll 80 eligible subjects with a target completion of 60 subjects. During the enrollment period, the subject drop-out rate with be closely monitored, if an unexpectedly high dropout rate is observed, then the targeted total enrollment number maybe be increased accordingly to ensure that a minimum of 60 subjects complete the study.

## 8.5. Statistical Significance Level

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 8.6. Handling of Missing Data and Drop-outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using fully Bayesian imputation by imputing missing values.

### 9. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

There will be no interim read performed on this study.

### 10. SUBJECT INFORMATION

## **10.1.** Disposition Information

Enrolled subjects will be allocated to one of the three mutually exclusive:

1. Completed: Subjects are considered to have completed the study if they (a) provided informed consent and/or assent; (b) they are eligible; (c) completed all three phases of testing; and (d) have not withdrawn/discontinued from the study.

- 2. Discontinued: Subjects are considered to have discontinued from the study if (i) test article was administered and (ii) discontinued from the study. Reasons for discontinuation include: (a) Adverse Event (b) unsatisfactory visual response due to test article (c) satisfaction lens fitting due to test article (d) lens discomfort (e) lens handling difficulties (e) withdrew consent during study (f) lost to follow-up (g) subject no longer meets eligibility criteria (h) subject withdrawn by PI to non-compliance to protocol (i) test article no longer available
- 3. Assigned and Test Article Administered: Total number subjects for which test articles were administered (Completed + Discontinued).
- 4. Enrolled but Not Dispensed: Subjects are considered to be Enrolled Not Dispensed Subjects if they were (i) enrolled to the study (provided informed consent and/or assent) but failed to satisfy the eligibility criteria (inclusion/exclusion criteria) or (ii) if they are randomized but did not receive a test article.
- 5. Total enrolled: Completed + Discontinued + Enrolled but Not Dispensed.

## 10.2. Protocol Deviations

Any protocol deviation that could impact the primary endpoints will result in the subject being excluded from the Per-Protocol analysis population. No analysis on protocol deviations will be performed. All reported protocol deviations will be listed.

# 10.3. Demographics and Baseline Characteristics

Demographic characteristics will be summarized by Per-Protocol, safety, and all enrolled population by strata (myopes and hyperopes) using descriptive statistics for continuous variables, and numbers and percentages of subjects for categorical variables. Demographic information will include age, gender, race, ethnicity and ADD power.

# 10.4. Treatment Compliance and Extent of Exposure

Average daily wear time and average daily comfort wear time will be provided in the summary table. Non-compliance will be reported in protocol deviation.

#### 10.5. Prior and Concomitant Medications

Prior and concomitant medications will be documented during screening and updated during the study when applicable. A listing for both prior and concomitant medications will be created for all enrolled subjects.

Disallowed medications for this study include: Anticholinergics, Oral Phenothiazines, Oral Retinoids, Corticosteroids and Oral Tetracycline.

Concomitant therapies that are disallowed include: Not applicable.

# 10.6. Medical History

A listing of medical and surgical history will be created for all enrolled subjects.

#### 11. STATISTICAL ANALYSIS

## 11.1. Primary Analysis

## **Primary Safety Analyses**

## **Strategy of Incorporating Historical Data:**

Safety analysis will be performed by incorporating of historical data from studies:

All these studies evaluated the same Test lens that was built in different manufacturing platforms to the same in vitro product requirements and are also considered to be representative of final commercial production. The historical individual data will be incorporated using is the power prior distribution (Ibrahim and Chen; 2000)<sup>3</sup>.

Let (y, z) and  $(y_0, z_0)$  denote the data from current study, and from historical data respectively, p the proportion of eyes with response 1 and  $\rho$  the correlation between left and right eyes. To construct a power prior distribution for parameter of interests  $(p, \rho)$ , we use the formula

$$P(p, \rho \mid y_0, z_0, a_0) \propto L(p, \rho \mid y_0, z_0)^{a_0} \pi_0(p, \rho),$$

where L(p,  $\rho \mid \mathbf{y_0}, \mathbf{z_0} \mid \mathbf{p}, \mathbf{p_0}$ )  $\propto P(\mathbf{y_0}, \mathbf{z_0} \mid \mathbf{p}, \rho)$  is the likelihood of (p,  $\rho$ ) based on the historical data and  $a_0$  is a discounting parameter constrained between 0 and 1. This parameter  $a_0$  controls the amount of the historical data we are borrowing:  $a_0 = 0$  corresponds to no incorporation of the historical data, while  $a_0 = 1$  corresponds to full borrowing of historical data. We set  $a_0 = 0.30$  for historical data of the Test lens was made in FMP and TAM21 platforms and  $a_0 = 0.10$  for Test lens made in the pilot line.

The posterior distribution of  $(p, \rho)$  given the current and historical data is

$$P(p, \rho | y, z, y_0, z_0, a_0) \propto L(p, \rho | y, z)L(p, \rho | y_0, z_0)^{a_0} \pi_0(p, \rho),$$

where  $L(p, \rho \mid y, z) \propto P(y, z \mid p, \rho)$  is the likelihood of  $(p, \rho)$  based on the current data.

#### **Primary Safety Analyses:**

Slit lamp finding grade 3 or higher and unacceptable lens fitting responses (yes/no) will be analyzed separately on the safety population using the Bayesian model described below. A sensitivity analysis will be conducted with no borrowing of historical data.

#### The Model:

Let Y1 and Y2 denote the binary outcomes for the left and right eyes, respectively, when wearing the test lens. Considering the correlation, ρ, between Y1 and Y2, the distribution of the CR-6400, Statistical Analysis Plan Version 1.0

sum Y = Y1 + Y2 is obtained by the mixture of two variables. One of them follow a binomial distribution Bin(2, p) with mixing probability (1- $\rho$ ) and the other one follows a modified Bernoulli distribution MBern(p), taking value 0 and 2 rather than conventional 0 and 1, with mixing probability p:

$$P(Y=y|\;p,\;\rho)=(1\text{-}\;\rho)Bin(2,\;p)I_{A1}+\;\rho MBern(p)I_{A2};$$
 where  $I_{A1}=\{0,\;1,\;2\}$  and  $I_{A2}=\{0,\;2\}$ 

To overcome the complexity of the mixture likelihood a latent variable  $Z_i$ , i = 1, 2 is introduced in the model to indicate in which component of the model the observation  $y_i$ , i=1, 2, belongs to, that is,

$$z_i = \begin{cases} 1, & \text{if the observation belong to the MBern(p),} \\ 0, & \text{if the observation belong to the Bin(2, p)} \end{cases}$$

The joint distribution of the augmented data (Y<sub>i</sub>, Z<sub>i</sub>), i=1, 2, is given by

$$P(Y = y_i, Z = z_i | p, \rho) = \rho^{z_i} p^{y_i z_i/2} (1 - p)^{(2 - y_i) z_i/2} (1 - \rho)^{1 - z_i} {2 \choose y_i} p^{y_i (1 - z_i)} (1 - p)^{(2 - y_i)(1 - z_i)}$$

The posterior distribution of  $(p, \rho)$  given (y, z),  $(y_0, z_0)$  and  $a_0$  is

$$P(p, \rho \mid | y, z, y_0, z_0, a_0) = P(y, z \mid p, \rho) P(y_0, z_0 \mid p, \rho)^{a_0} \pi_0(p, \rho)$$

where,  $\pi_0$  is joint prior distribution of  $(p, \rho)$ . Here we assume p and  $\rho$  to be independent with a prior beta  $(\alpha, \beta)$  for p and uniform (0,1) for  $\rho$ . Hence the joint distribution of  $(p, \rho)$  is given by  $\pi_0$   $(p, \rho | \alpha, \beta) \propto p^{\alpha-1}(1-p)^{\beta-1}$ . The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC Procedure will be used to estimate the posterior distributions of the parameters  $(p, \rho)$ . Inferences will be made based on a posterior credible interval for the relevant parameters.

### **Hypothesis Testing**

With respect to unacceptable lens fit the null and alternative hypothesis for superiority is as follows:

$$H_o: p_T \ge 0.05$$
  
 $H_A: p_T < 0.05$ 

Where,  $p_T$  represents the proportion of subject eyes that are considered to have unacceptable fit for the study lens after 2-weeks of lens wear. Success for unacceptable fit will be declared if the upper bound of the 2-sided 95% credible interval of the proportion is lower than 0.05; i.e.  $P(p_T < 0.05) \ge .975$ .

With respect to Grade 3 or Higher SLFs the null and alternative hypothesis for superiority is as follows:

$$H_o: p_T \ge 0.05$$

$$H_A: p_T < 0.05$$

Where,  $p_T$  represents the proportion of subject that experienced any Grade 3 or Higher SLF or experienced a corneal infiltrate. Success for Grade 3 or higher SLFs will be declared if the upper bound of the 2-sided 95% credible interval of the proportion is lower than 0.05; i.e.  $P(p_T < 0.05) \ge .975$ .

If no SLF findings of Grade 3 or higher or unacceptable lens fit is observed, alternative analysis methods may be considered.

# **Primary Efficacy Analyses**

Efficacy analysis will be conducted the Per-Protocol Population without borrowing from historical data. A sensitivity analysis will be performed by incorporating historical data. The level of borrowing used in the safety analysis will be considered. Further sensitivity analyses on the Safety population may also be considered if the observed subject dropout rate exceeds 15%.

#### **CLUE Vision**

CLUE vision scores will be analyzed using a multivariate Bayesian normal random effects model. The model will include baseline clue score, age, add power, gender and strata (Hyperopes and Myopes) as fixed effects. Site will be included as a random effect. An unstructured (UN) covariance structure will be used to model the residual errors from measurements within the same subject across timepoints. Heterogeneous residuals covariance structures (R-side) across strata will be considered when appropriate.

#### The Model:

Let  $y_{ijk} = (y1_{ijk}, y2_{ijk})^T$  denote the CLUE vision scores for the  $K^{th}$  subject at the  $J^{th}$  site, in  $i^{th}$  stratum (Hyperope or Myope) at the 3-Day and 2-Week Follow-up evaluations. The likelihood for  $y_{ijk}$  is constructed as follows:

$$y_{iik} \sim N(\mu_{iik}, \Sigma)$$

 $\mu_{ijk} = (\mu 1_{ijk}, \mu 2_{ijk})^T$  and  $\Sigma$  is a 2X2 variance-covariance matrix. Here,

$$\begin{array}{lll} \mu \mathbf{1}_{ijk} = & \pi_1 + \ \mu_0 + \ \beta_1 Baseline_k + \beta_2 age_k + \ \beta_3 stratum_k + \beta_4 Gender_k + \beta_5 ADD_k + \ \gamma_j \\ \mu \mathbf{2}_{ijk} = & \pi_2 + \ \mu_0 + \ \beta_1 Baseline_k + \beta_2 age_k + \ \beta_3 stratum_k + \beta_4 Gender_k + \beta_5 ADD_k + \ \gamma_j \\ \end{array}$$

In this model  $\pi_1$ ,  $\pi_2$ , represent the effect of time point with the constraint  $\pi_1 + \pi_2 = 0$ . In this model, we define  $stratum_k = 0$  for the Myope Strata and  $stratum_k = 1$  for the Hyperope Strata. So  $\beta_3$  stands for the difference between the Hyperope and Myope Strata with respect to CLUE vision; A positive  $\beta_3$  indicates the Hyperopes performed better than the Myopes.

We assume random site effects are independent and identically distributed (i.i.d) as  $\gamma_j \sim N(0, \sigma_{site}^2)$  for site for j=1, 2, 3, 4, 5..., 11 (site). For the  $\beta$  coefficients, independent non-informative **CR-6400**, Statistical Analysis Plan Version 1.0

priors N(0, 1000) will be used. For the variance of random effect of  $\sigma_{site}^2$  an independent non-informative conjugate prior, inverse-gamma(0.001, 0.001) will be used. For  $\Sigma$ , non-informative conjugate priors inverse-Wishart(2,S) will be used where S is a 2X2 variance-covariance matrix of  $y_{ijk}$ . The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC 15.15 procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

## **Hypothesis Testing**

Hypothesis testing for CLUE Vision Scores endpoints will be conducted separately for each stratum (Hyperope and Myope):

The null and alternative hypotheses for CLUE vision for statistical superiority of the Hyperope stratum are as follows:

$$H_o: \mu_{Hyperope} \leq 32$$

$$H_A$$
:  $\mu_{Hyperope} > 32$ 

The null hypothesis will be rejected if the lower bound of the 2-sided 95% credible interval of the clue vision posterior mean estimate for the Hyperope stratum is above 32. i.e.,  $P(\mu_{Hyperopes} > 32) > 0.975$ .

The null and alternative hypotheses for CLUE vision for statistical superiority of the Myopes stratum are as follows:

$$H_o$$
:  $\mu_{Mvove} \le 40$ 

$$H_A$$
:  $\mu_{Myope} > 40$ 

The null hypothesis will be rejected if the lower bound of the 2-sided 95% credible interval of the clue vision posterior mean estimate for the Myope stratum is above 40. i.e.,  $P(\mu_{Myopes} > 40) \ge 0.975$ .

#### Binocular Visual Performance

Binocular high luminance, high contrast (HLHC) visual performance (logMAR) at the 2-week follow-up evaluation will be analyzed using a Bayesian normal random-effects model for repeated measures. The model will include strata (Hyperope and Myope), add power, age, gender as fixed effects. Site and will be included as a random effect. An unstructured (UN) covariance structure will be used to model the residual errors from measurements within the same subject across different positions. Heterogeneous residuals covariance structures (R-side) across position will be considered when appropriate.

Let  $y_{ijkl}$  denote the visual performance for the study lens for the  $j^{th}$  subject in the  $k^{th}$  strata (Hyperope or Myope), at the  $l^{th}$  site for the  $i^{th}$  position.

The Model:

 $y_{ijkl} = \mu_0 + \beta_1 \ age_i + \beta_2 \ addpwr_j + \beta_3 \text{dist\_yn} \ _i + \beta_4 \text{inter\_yn} \ _i + \beta_5 Female_j + \beta_6 Strata_k \ _+ \delta_l + \varepsilon_{ijkl}$ 

- $\mu_0$ : overall intercept
- $addpwr_i$ : ADD Power
- dist\_yn k: Distance vs. Intermediate and Near
- inter\_yn k: Intermediate vs. Distance and Near
- Female<sub>i</sub>: Female indicator; Female=1 if sex='Female' and 0 otherwise
- Strata<sub>i</sub>: Strata indicator; Strata=1 if strata='Hyperope' and 0 otherwise
- $\delta_l$ : effect of the  $l^{th}$  clinical site, a random effect
- $\varepsilon_{jkl}$ : random error associated with the  $i^{th}$  position for the  $j^{th}$  subject in the  $k^{th}$  strata at the  $l^{th}$  investigational site

Here we assume  $\delta_i$  and  $\varepsilon_{ikl}$  are independent where

$$\bullet \quad \delta_{j} \sim N(0, \sigma_{site}^{2}) ;$$

$$\bullet \quad \begin{bmatrix} \varepsilon_{1jkl} \\ \varepsilon_{2jkl} \\ \varepsilon_{3jkl} \end{bmatrix} \sim N \begin{pmatrix} \begin{bmatrix} 0 \\ 0 \\ 0 \end{bmatrix}, \begin{bmatrix} \sigma_{11}^{2} & \sigma_{12} & \sigma_{13} \\ \sigma_{21} & \sigma_{22}^{2} & \sigma_{23} \\ \sigma_{31} & \sigma_{32} & \sigma_{33}^{2} \end{bmatrix} \end{pmatrix}$$

We assume random site effects are independent and identically distributed (i.i.d) as  $\gamma_j \sim N(0, \sigma_{site}^2)$  for site for j=1, 2, 3, 4, 5..., 11 (site). For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effect of  $\sigma_{site}^2$  an independent non-informative conjugate prior, inverse-gamma(0.001, 0.001) will be used. For the variance of  $y_{ijkl}$  an independent non-informative conjugate prior, inverse-gamma(0.001, 0.001) will be also used. The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC 15.1<sup>5</sup> procedure will be used to estimate the posterior distribution of the unknown parameters. Inferences will be made based on the 95% posterior credible intervals for relevant parameters.

### **Hypothesis Testing**

The null and alternative hypothesis for binocular distance HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.10 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.10 \log MAR$ 

Superiority will be declared if the upper limit of the 95% CrI is below 0.10 logMAR. i.e.  $P(\mu_{Test} < 0.10) \ge 0.975$ .

The null and alternative hypothesis for binocular near HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Superiority will be declared if the upper limit of the 95% CrI is below 0.17 logMAR. i.e.  $P(\mu_{Test} < 0.17) \ge 0.975$ .

The null and alternative hypothesis for binocular distance HLHC visual performance to test for superiority of the Test lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Superiority will be declared if the upper limit of the 95% CrI is below 0.17 logMAR. i.e.  $P(\mu_{Test} < 0.17) \ge 0.975$ .

## 11.2. Secondary Analysis

Proportion of Subjects with Optimal Lens Pair

The number of lenses used for each subject will be calculated as the original pair (2) plus all the required modifications to reach the optimal pair. In this study the minimum number of lenses per subject used would be 2 where the max would be 6. The data will be dichotomized as 1 if the subject was able to achieve optimal lens pair in 4 lenses or less and 0 otherwise. The binary response will be analyzed using Bayesian logistic regression random-effects model to estimate the proportion of eyes that reached optimal lens pair in 4 lenses or less. The regression model will include strata (Hyperope and Myope), add power, age, gender, event (fitting, optimization, 2-week follow-up) and the interaction between strata by event. Site will be included in the model as a random effect. Non-informative priors will be used for the unknown parameter. For the  $\beta$  coefficients, independent non-informative priors N(0, 1000) will be used. For the variance of random effects of  $\sigma_{\text{site}}^2$  non-informative conjugate prior, inverse-gamma (0.001, 0.001) will be used. Inferences will be made based on the posterior credible interval for the relevant parameters.

## **Hypothesis Testing**

With respect to the proportion of subjects that have achieved optimal fitting in 4 lenses or less, the null and alternative hypothesis for superiority is as follows:

$$H_o: p_T \le 0.90$$
  
 $H_A: p_T > 0.90$ 

Where,  $p_T$  represents the proportion of subjects that have achieved optimal fitting in 4 lenses or less. Success for will be declared if the lower bound of the 2-sided 95% credible interval of the proportion is greater than 0.90; i.e.  $P(p_T > 0.90) \ge .975$ .

If not enough events occur during the duration of this study the model presented for the safety population.

## 11.3. Other Analysis

There are no other pre-planned analyses for this study.

### 12. SAFETY EVALUATION

#### 12.1. Adverse Events

Listings of all reported ocular and non-ocular AEs and SAEs will be reported and will include lens type, eye diagnosis, severity of the AE, the number of days the subject spent in the study, the slit lamp findings at discovery of the AE, whether or not it is lens related, the possible cause, and treatments provided to the patient, the outcome, the subjects final Snellen visual acuity, whether or not the subject eye had a scar at the resolution of the AE and the action taken. In addition, the total number of subjects and the total number of eyes with each type of AE (SAEs, ocular AEs and non-ocular AEs) will be tabulated and presented as a footnote in each summary.

# 12.2. Keratometry and Over Refraction

Keratometry will be assessed for each eye at Entrance (Visit 1) for the following metrics: (1) Steep Dioptric Power, (2) Steep Degrees, (3) Flat Dioptric Power and (4) Flat Degree. Each keratometry metric will be summarized using n, mean, min, and max across eye type and summarized by stratum (Hyperopes and Myopes) and across all subjects.

## 12.3. Contact lens Corrected Visual Acuity

Contact lens visual acuity will be assessed using Snellen visual acuity Charts at both 4m (Distance) and 40cm (Near) at the fitting evaluation, lens dispensing, 3-day follow-up and the 2-week Follow-up evaluations. CLVA will be assessed both monocularly and binocularly. Summaries for Monocular CLVA and binocular CLVA will be presented using counts and percentages of eyes and subjects, for monocular CLVA and binocular CLVA, respectively.

#### 12.4. Reasons for Discontinuation

The number of discontinued subjects by the analysis time point will be displayed by visit. Reasons for discontinuation include the following:

- 1. Adverse Event
- 2. Unsatisfactory lens fitting due to test article
- 3. Unsatisfactory visual response due to test articles

- 4. Lens discomfort
- 5. Withdrew consent during study
- 6. Lost to follow-up
- 7. Subject no longer meet eligibility criteria
- 8. Subject withdrawn by PI due to non-compliance to protocol
- 9. Test article no longer available
- 10. Other

## 12.5. Unscheduled Lens Replacement

The number of unscheduled lens replacements and corresponding reasons will be tabulated by visit and overall, across eyes for both completed and discontinued eyes.

# 12.6. Physical Examination Findings

Slit lamp findings will be assessed for each subject eye at baseline, 3-day Follow-up, the 2-week follow-up and at any unscheduled visit using the FDA Grading scale (Grade 0=None, Grade 1=Trace, Grade2=Mild, Grade 3=Moderate, Grade 4=Severe). Slit lamp finding assessments include the following metrics:

- Corneal Infiltrates (Yes/No)
- Corneal Edema
- Corneal Neovascularization
- Corneal Neovascularization Location
- Corneal Staining
- Corneal Staining Location
- Conjunctival Injection
- Tarsal Abnormalities
- Other

# 12.7. Clinical Laboratory Tests

Not applicable.

# 12.8. Other Safety Parameters

#### Subject's Reported Ocular Symptoms

Frequency and severity by eye of subject's reported ocular symptoms and problems with the study lens at fitting and post-fitting evaluation visits including the 2-Week Follow-up and unscheduled visits. Severity of the symptoms can be:

- 0 = Not Applicable or Not Recorded;
- 1 = Mild and results in little or no interference with lens wear;
- 2 = Moderate AND/OR occasionally interferes with lens wear;
- 3 = Severe AND/OR frequently interferes with lens wear.

#### Lens fitting characteristics

Frequency by eye of mechanical lens fitting characteristics at fitting and 2-Week Follow-up evaluations. Lens fitting characteristics to be reported are:

- Lens Centration Grade
- Decentered Direction
- Limbal Exposure Grade
- Edge Lift (Present or Absent)
- Primary Gaze Movement Grade
- Upgaze Movement Grade
- Lens Tightness Grade (Push-up Test)
- Acceptable Fitting (yes/no)

## Contact Lens Deposits

Contact lens deposits will be assessed for each eye at the 2-week Follow-up on the front and back surface of the study lens; the amount of deposits will be Graded using the scale:

- None = Grade 0 (No deposition).
- Slight = Grade 1 (Deposition which occupies 1-5% of the lens surface area.)
- Mild = Grade 2 (Deposition which occupies 6-15% of the lens surface area.)
- Moderate = Grade 3 (Deposition which occupies 16-25% of the lens surface area.)
- Severe = Grade 4 (Deposition which occupies =26% of the lens surface area.)

## Contact Lens Wettability

Contact lens Wettability will be assessed for each eye at the 2-week Follow-up. Wettability will be Graded using the scale:

- Grade 0 = All regions of lens surface are wettable between blinks (a minimum of 6 seconds between blinks).
- Grade 1 = Discrete non-wetting area(s) after a minimum of 3 seconds post blink.
- Grade 2 = Single non-wetting area within 2-3 seconds of blink.
- Grade 3 = Several non-wetting areas within 2-3 seconds of blink.
- Grade 4 = Immediate area(s) of non-wetting after blink.

## 13. REFERENCES

- 1. Wirth RJ, et al. Development of the Contact Lens User Experience: CLUE Scales. Optom Vis Sci. 2016; 93(8): 801-808.
- 2. SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC: SAS Institute Inc; 2014.
- 3. Ibrahim JG, Chen M-H, Gwon Y, Chen F. The power prior: theory and applications. Stat Med. 2015;34(28):3724-3749.
- 4. Jovanovic, B.D. and Levy, P.S. (1997). A Look at the Rule of Three. *The American Statistician* **51**, 137-139.
- 5. SAS Institute Inc. 2018. SAS/STAT® 15.1 User's Guide. Cary, NC: SAS Institute Inc.

# 14. APPENDICES

# 14.1. Time and Event Schedule

| Visit Information | Visit 1 Screening, Baseline, Treatment 1 Fitting | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3<br>Treatment 1<br>Follow-up 2 |
|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 12±2<br>from V2 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours |
| Statement of Informed | | | |
| Consent | X | | |
| Demographics | X | | |
| Medical | | | |
| History/Concomitant | | | |
| Medications | X | | |
| Adverse Events and | | | |
| Concomitant | | | |
| Medications Review | | X | X |
| Compliance | | X | X |
| Habitual Contact Lens | | | |
| Information | X | | |
| Contact Lens History | X | | |
| Wear Time and | | 3 | |
| Comfortable Wear | | | |
| Time with Habitual | | | |
| Lenses | X | | |
| Wear Time and | | 2 | |
| Comfortable Wear | | | |
| Time with Study | | | |
| Lenses | | X | X |
| Screening | | | |
| Inclusion/Exclusion | | | |
| Criteria | X | | |
| Subject Reported | | | |
| Ocular Symptoms | X | X | X |
| Baseline | | | |
| Questionnaire | X | | |
| CLDEQ-8 | | | |
| Questionnaire | X | X | X |

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| VISIT IIIIOIIIIAIIOII | Screening, | Treatment 1 | Treatment 1 |
| | 900 | | |
| | Baseline, | Follow-up 1 | Follow-up 2 |
| | Treatment 1 | Optimization | |
| T. D. | Fitting | D 211 | D 1010 |
| Time Point | Day 0 | Day 3±1 | Day 12±2 |
| | 0.51 | from V1 | from V2 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours |
| Distance and Near | | | |
| Entrance Visual | | | |
| Acuity | X | X | X |
| Lens Removal | X | X | X |
| Keratometry | X | | |
| Subjective Refraction | | | |
| and Distance Visual | | | |
| Acuity | X | | |
| Near ADD | | | |
| Determination | X | | |
| Ocular Dominance | X | | |
| ADD Refinement | X | | |
| Near Visual Acuity | X | | |
| Biomicroscopy | X | X | X |
| Baseline | | | |
| Inclusion/Exclusion | | | |
| Criteria | X | | |
| Eligibility | X | | |
| Lens Selection | X | x (if modified) | |
| Lens Insertion | X | X | X |
| 10 Minute Settling | X | x (if modified) | |
| Visual Satisfaction / | | | |
| Subjective Acceptance | X | X | X |
| Study Lens Distance | | | |
| and Near Visual | | | |
| Acuity | X | X | x |
| Distance Over | | 3 | - |
| Refraction and Visual | | | |
| Acuity | X | X | |
| Lens Fit Assessment | X | X | X |
| Binocular Over | one of the state o | - VIII-VI | 3100 |
| Refraction | | X | X |
| Lens Deposits | | | X |
| Lens Wettability | | | X |

CR-6400, Statistical Analysis Plan Version 1.0

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 |
| | Baseline, | Follow-up 1 | Follow-up 2 |
| | Treatment 1 | Optimization | |
| | Fitting | 30 | |
| Time Point | Day 0 | Day 3±1 | Day 12±2 |
| | -2/ | from V1 | from V2 |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours |
| Duration | | | |
| Visual Performance | | | X |
| Modifications | X | X | |
| Post-Fit GSI | | | |
| Questionnaire | X | X | |
| Worn Lens Collection | | x | x |
| Study Lens | | | |
| Questionnaire | | X | X |
| Distance and Near | | | |
| Exit Visual Acuity | X | X | |
| Dispensing Criteria | X | X | |
| Instructions | X | X | |
| Schedule Follow-up | X | X | |
| Final Evaluation | | | X<br>(or when subject<br>discontinued) |

## 14.2. Statistical Analysis Code

## 14.2.1. Primary Analysis

**CLUE Vision** 

```
PROC MCMC DATA =ads NTHREADS =12 SEED =18965237 NBI =15000 NMC
=100000 THIN=20 DIAG = ALL OUTPOST = simout DIC PLOTS(SMOOTH FRINGE) =
ALL MCHISTORY = BRIEF PROPCOV = QUANEW STATS = ALL STATS(ALPHA =
(0.05) PERCENTAGE = (2.5 50 97.5)) plots(smooth)=ALL MONITOR=( parms
Hyperopes 3day Myopes 3day Hyperopes 2wk Myopes 2wk);
ARRAY aval[2] FU1 FU2;
ARRAY mu[2] mu1 mu2;
ARRAY sigma[2,2];
ARRAY S[2,2] (10)
            01);
PARMS p1 0.5 p2 0.1 beta0-beta5;
PARMS sigma { 1 0
             0 1};
PARMS sigma_site;
            \sim NORMAL(0, var = 1000);
PRIOR beta:
prior p: ~ NORMAL(0, var=1000);
PRIOR sigma
             \sim IWISH(2, S);
PRIOR sigma site \sim IGAMMA(shape = 0.01, scale = 0.01);
RANDOM gamma site ~ NORMAL(0, VAR = sigma site) SUBJECT = siteid;
mu1 = p1 + beta0 + beta1*stratan + beta2*Base + beta3*age + beta4*sexn + beta5*addpwr +
Gamma site;
mu2 = p1 - p2 + beta0 + beta1*stratan + beta2*Base + beta3*age + beta4*sexn + beta5*addpwr
+ Gamma site;
MODEL aval ~ MVN(mu, sigma);
 BEGINNODATA;
      Hyperopes 2wk = p1
                             + beta0 + beta1 + 0.5*beta4;
      Myopes 2wk = p1
                             + beta0 + 0.5*beta4;
      Hyperopes 3Day = p1 - p2 + beta0 + beta1 + 0.5*beta4;
      Myopes 3Day = p1 - p2 + beta0
                                          + 0.5*beta4;
 ENDNODATA;
RUN;
Where,
CR-6400, Statistical Analysis Plan Version 1.0
```

```
Ads = Analysis dataset for CLUE Vision Scores
Stratan=numerical representation of strata, where Hyperopes=1 and Myopes=0
Base= Baseline CLUE Vision Score
Age= Age of subject at time of consent
Sexn=numerical representation of sex, where Female=1 and Male=0;
Addpwr=Add power of subject at baseline
Siteid=Site Identifier
```

#### Visual Performance

```
PROC MCMC DATA =ads vp NTHREADS=12 SEED=20180906 NBI=80000 NMC=150000
THIN=30 DIAG=ALL OUTPOST=simout DIC PLOTS(SMOOTH FRINGE)=ALL
MCHISTORY=BRIEF PROPCOV=QUANEW STATS=ALL STATS(ALPHA = (0.05)
PERCENTAGE=(2.5 50 97.5)) plots(smooth)=ALL MONITOR=( parms mu D mu I
mu N);
PARMS beta 0 beta 1 0 beta 2 0 beta 3 0 beta 4 0 beta 5 0 beta 6 0;
PARMS s2 1;
PARMS s2g_site s2g_site1;
PRIOR beta: \sim NORMAL(0, var = 1000);
PRIOR s2 \sim IGAMMA(.001, s = .001);
PRIOR s2g site s2g subj~ IGAMMA(.001, s =.001);
RANDOM Gamma site \sim NORMAL(0, VAR = s2g site) SUBJECT=SITEID;
RANDOM Gamma subj ~ NORMAL(0, VAR = s2g subj) SUBJECT=USBJID;
mu = beta0 + beta1*dist yn + beta2*inter yn + beta3*age + beta4*sexn + beta5*stratan +
beta6*addpwr + Gamma subj + Gamma site;
MODEL AVAL \sim NORMAL (mu, VAR = s2);
BEGINNODATA;
   mu D = beta0 + beta1 + 0.5*beta4 + 0.5*beta5;
   mu I = beta0 + beta2 + 0.5*beta4 + 0.5*beta5;
  mu N = beta0
                     + 0.5*beta4 + 0.5*beta5;
ENDNODATA;
 RUN;
```

Where,

ads vp = Analysis dataset for Binocular HLHC Visual Performance dist\_yn= numerical representation of position, where distance=1 and Intermediate and Near=0

inter\_yn= numerical representation of position, where Intermediate=1 and Distance and Near=0 Stratan=numerical representation of strata, where Hyperopes=1 and Myopes=0

Age= Age of subject at time of consent Sexn=numerical representation of sex, where Female=1 and Male=0; Addpwr=Add power of subject at baseline Siteid=Site Identifier

## SLF (Grade 3 or Higher) and Unacceptable Lens Fitting

```
    With Borrowing

PROC MCMC DATA= ADS DIC =brief
NBI=50000 NMC=80000 THIN=15 STATS=ALL MONITOR=( parms )STATS(ALPHA=(0.05)
PERCENTAGE=(2.5 25 50 75 97.5) ) SEED=14789652 ;
PARM p ro .5;
PRIOR ro ~ UNIFORM(0,1);
PRIOR p \sim BETA(0.5, 0.5);
BEGINCNST;
IF studyid in \bigcirc ) THEN a0 = 0.3;
ELSE IF studyid in ( THEN a0 = 0.3;
ELSE IF studyid in
                                                                                                    ) THEN a0=0.1;
ENDCNST;
llike = log( (1-ro)*PDF('BINOMIAL', y, p, 2) + z*ro*(p**y*(1-p)**(2-p)**(1-p)**(2-p)**(1-p)
y)) ** (1/2));
IF studyid in ( THEN llike = llike; ELSE llike = a0*llike;
MODEL y ~ GENERAL(llike);
RUN;

    Without Borrowing

PROC MCMC DATA= ADS DIC =brief
NBI=50000 NMC=80000 THIN=15 STATS=ALL MONITOR=( parms )STATS(ALPHA=(0.05)
PERCENTAGE=(2.5 25 50 75 97.5) ) SEED=14256983 ;
PARM p ro .5;
PRIOR ro ~ UNIFORM(0,1);
PRIOR p \sim BETA(0.5, 0.5);
BEGINCNST;
IF studyid in (\mbox{\ \ ELSE\ IF\ } ) THEN a0 = 0; ELSE IF studyid in (\mbox{\ \ \ \ }) THEN a0 = 0;
ELSE IF studyid in
                                                                                                                                                                                 THEN a0=0;
ENDCNST;
llike = log( (1-ro)*PDF('BINOMIAL', y, p, 2) + z*ro*(p**y*(1-p)**(2-p)**(1-p)**(2-p)**(1-p)
\forall)) ** (1/2));
IF studyid in ( THEN llike = llike; ELSE llike = a0*llike;
MODEL y ~ GENERAL(llike);
RUN;
```

## Where,

ads = Analysis dataset for Grade 3 or higher SLFs or Unacceptable Lens Fitting a0 = degree of borrowing stuyid=Study Identifier